CLINICAL TRIAL: NCT03419832
Title: The NEAT Study: An Examination of a Novel Consent Form Design in a Real-world Setting
Brief Title: The New Executive and Appendix Template (NEAT) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00031904; 5UL1TR001420-03 (NIH)
Record Dates: First submitted 2018-01-22; First posted 2018-02-05 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Comprehension; Informed Consent
Keywords: ARIC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEAT Form (Experimental): Study participants will be randomized to the NEAT form and the materials that accompany it (also detailing the ARIC study).
  Interventions: Other: NEAT Form
- Standard Form (Active Comparator): Study participants will be randomized to the traditional standard consent form (detailing the ARIC study).
  Interventions: Other: Standard Form

INTERVENTIONS:
Other: NEAT Form — The NEAT form consists of a clear and concise overview document containing information satisfying all elements of consent. This is made up of IRB-approved wording from the regular consent form. More detailed information, such as specific clinic measures are provided as additional material and are discussed during the consent process after the general overview has been provided with the NEAT form.
  Arms: NEAT Form
Other: Standard Form — The regular IRB approved version.
  Arms: Standard Form

SUMMARY:
There is evidence that the current design and content provided by most biomedical research informed consent documents do not consistently meet the expectations researchers place on them to effectively inform research participants of information thought to be most important in facilitating their ability to make informed decisions about participation. The need for revisions to the informed consent document design is supported by empirical research.This pilot study will examine the effectiveness of the New Executive and Appendix Template (NEAT) form when used in the consent process for individuals participating in the Atherosclerosis Risk in Communities (ARIC) Neurocognitive Study.

DETAILED DESCRIPTION:
The importance of informed consent is to ensure that participants in clinical research are provided the opportunity to make autonomous choices is a paramount ethical premise in human research. The effectiveness of consent document design and consent process to accurately and fully convey the elements of informed consent is critical and deserves further study. Development of an improved informed consent document design for clinical studies would be a valuable contribution to human research. Chunking sentences or phrases in text into related groupings resulted in a positive significant improvement in reading comprehension among students with poor reading skills. Because the information contained in consent documents can be complex, detailed, and novel for potential research participants, the use of a modified form of chunking may be an effective and a low cost way of improving comprehension of the elements of consent. Specifically, the primary objective of the study is to determine if participants who receive the NEAT form report greater comprehension at the end of the consent process, than participants who receive a standard form.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are eligible for the ARIC study, with which this pilot study is cooperating.

Exclusion Criteria:

* Any individuals not eligible for the ARIC study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Andrews, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NEAT Form | Standard Form
Started | 52 | 49
Completed | 52 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Data was not collected except to confirm that subjects were 65 or older.
Groups:
- Total: Total of all reporting groups
Arm/Group | NEAT Form | Standard Form | Total
Number analyzed (Participants) | 52 | 49 | 101
Age, Customized [Count of Participants; unit: Participants] — Specific age was not collected. The study team only confirmed that participants were 65 or older.
  Participants
    Aged 65 or older | 52 | 49 | 101
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender baseline characteristic data was not collected for this study.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Comprehension of the NEAT Form
Description: Following the consent process, participants will be administered the Comprehension tool to measure their comprehension. The summary scores will be used to address the primary aim of whether or not the NEAT consent form improves participant comprehension. There are 7 questions, each question is rated 0-2 with a total scale of 0-14. Higher values denotes better outcomes.
Time Frame: at visit one, up to 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NEAT Form | Standard Form
Number analyzed (Participants) | 52 | 49
score on a scale | 10.6 (2.1) | 10.2 (2.5)

2. Secondary Outcome: Qualitative Analysis of the Readability and Understandability of the Consent Form by Participants
Description: Subjects were asked about the readability and understandability of the consent form and selected responses from the following options: Much easier to read and understand, Somewhat easier to read and understand, About the same, or Harder/Much harder to read and understand. The frequency of each response was reported.
Time Frame: at visit one, up to 24 hours
Population: Two people did not complete this question in the Standard Form Arm
Measure: Number; unit: number of each response
Arm/Group | NEAT Form | Standard Form
Number analyzed (Participants) | 52 | 47
number of each response
  Much easier to read and understand | 18 | 9
  Somewhat easier to read and understand | 12 | 9
  About the same | 19 | 24
  Harder/Much harder to read and understandBottom of Form | 3 | 5

3. Secondary Outcome: Qualitative Analysis of the Format and Design of the Consent Form by Participants
Description: Subjects were asked about the format and design of the consent form and selected from the following options: Much better format and design, Somewhat better format and design, About the same format and design, or Somewhat worse format and design. The frequency of each response was reported.
Time Frame: at visit one, up to 24 hours
Population: Two people did not complete this question in the Standard Form Arm.
Measure: Number; unit: number of each response
Arm/Group | NEAT Form | Standard Form
Number analyzed (Participants) | 52 | 47
number of each response
  Much better format and design | 14 | 13
  Somewhat better format and design | 22 | 14
  About the same format and design | 16 | 18
  Somewhat worse format and design | 0 | 2

4. Secondary Outcome: Qualitative Analysis of the Time of Discussion of the Consent Form by Participants
Description: Subjects were asked about the time of discussion of the consent form and selected from following options: Much shorter time, Somewhat shorter time, About the same time, or Somewhat/Much longer time. The frequency of each response was reported.
Time Frame: at visit one, up to 24 hours
Population: Two people did not complete this question in the Standard Form Arm.
Measure: Number; unit: number of each response
Arm/Group | NEAT Form | Standard Form
Number analyzed (Participants) | 52 | 47
number of each response
  Much shorter time | 9 | 9
  Somewhat shorter time | 16 | 9
  About the same time | 18 | 13
  Somewhat/Much longer time | 9 | 16

5. Secondary Outcome: Qualitative Analysis of the Format and Design of the Consent Form by Study Team
Description: The study team member qualitative data about their opinion of using the form will be collected. Study team members were asked about the format and design of the consent form and selected from the following options: Much better format and design, Somewhat better format and design, About the same format and design, or Somewhat worse format and design. The frequency of each response was reported.
Time Frame: at visit one, up to 24 hours
Population: Data not collected for this outcome. No data to report.
Arm/Group | NEAT Form | Standard Form
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: from time of consent through end of study, up to 24 hours
Arm/Group | NEAT Form | Standard Form
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49
Other Adverse Events (participants affected / at risk) | 0/52 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT03419832/Prot_SAP_000.pdf